CLINICAL TRIAL: NCT01457859
Title: Effectiveness of Triclosan Coated VICRYL\MONOCRYL Sutures in Preventing Leg Wound Infection Compared to POLYSORB\ BIOSYN Sutures in Patients After Coronary Bypass Surgery- a Randomized Controlled Trial
Brief Title: Effectiveness of Triclosan Coated Sutures in Preventing Leg Wound Infection After Coronary Artery Bypass Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Dr. Shani Liran, Cardiac surgery resident, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RMB-0228.CTIL
Record Dates: First submitted 2011-10-16; First posted 2011-10-24 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Complication of Coronary Artery Bypass Graft; Surgical Wound Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Triclosan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional sutures (Active Comparator)
  Interventions: Other: Conventional non-coated surgical sutures
- Antiseptic sutures (Experimental)
  Interventions: Drug: Triclosan

INTERVENTIONS:
Drug: Triclosan — Triclosan coated surgical sewing threads (VICRYL+ and MONOCRYL+) applied for leg wound closure after CABG
  Arms: Antiseptic sutures
Other: Conventional non-coated surgical sutures — Conventional non-coated surgical sewing threads (POLYSORB and BIOSYN) will be applied after CABG for leg wound closure
  Arms: Conventional sutures

SUMMARY:
The purpose of this study is to assess whether triclosan-coated sutures reduces wound infections compared to regular non-coated sutures, after saphenous vein harvesting in CABG patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older with written informed consent
* Male and female subjects
* Subjects scheduled for an elective and urgent CABG surgery that includes saphenous vein harvesting.

Exclusion Criteria:

* Known allergy or intolerance to triclosan
* Different surgical prophylactic antibiotic regimen than common in the department.
* Continuous preoperative and predicted postoperative antibiotic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
leg wound infection | Up to 45 days postsurgery
  Proportion of subjects with leg wound infection in research versus control group within 45 days of surgery according to CDC SSI criteria

SECONDARY OUTCOMES:
Antibiotics administration | Up to 45 days postsurgery
  Amount of administered antibiotic for leg wound infection after surgery
Hospital Length of stay | Average of 7 days postsurgery
Incidence of hospital re-admission due to leg wound infection | Within 45 days postsurgery

CONTACTS AND LOCATIONS:
Overall Officials: Liran Shani, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Depatment of cardiac surgery, Haifa, Israel